CLINICAL TRIAL: NCT06377644
Title: Comparing the Efficacy of Kinesology Taping Versus Dry Needling With Conventional Treatment for Improving Quality of Life and Alleviating Pain in Frozen Shoulder Patients
Brief Title: Comparing the Efficacy of KT vs DN With Conventional Treatment for Improving QOL and Alleviating Pain in Frozen Shoulder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall19/560
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling (Other)
  Interventions: Diagnostic Test: Dry Needling
- Kinesio taping (Experimental)
  Interventions: Diagnostic Test: Kinesio taping

INTERVENTIONS:
Diagnostic Test: Kinesio taping — Kinesio taping is a physiotherapy method employed to provide support and stability to muscles and joints while allowing freedom of movement (ROM). The elastic nature of kinesio tape closely resembles that of human skin. After application, kinesio tape rebounds, generating a pulling force that acts as the primary stabilizer for the specific area. Physiotherapy treatments often involve a combination of stretching and strengthening exercises, along with electrotherapy modalities. Additionally, Joint mobilization is a form of passive movement in a broad spectrum of exercise used to treat painful and stiff synovial joints.
  Arms: Kinesio taping
Diagnostic Test: Dry Needling — Dry needling is a minimally invasive technique involving the use of a single filament or acupuncture needle to penetrate painful soft tissue areas. From a neurophysiological standpoint, Dry Needling might stimulate A-delta nerve fibers (group III), which could activate inhibitory dorsal horn interneurons containing enkephalin, leading to pain suppression and relief through opioid mechanisms. (DN) may affect microcirculation. Numerous studies have shown that inserting needles into muscles can increase blood flow in both the skin and the muscle in the treated area. It can lead to an immediate reduction in local and referred pains, as well as enhance range of motion (ROM) and correct muscle activity patterns.
  Arms: Dry Needling

SUMMARY:
"Randomized control trial is our study design, we will make 2 groups group A ( 15 patients of frozen shoulder) and Group B (15 patients of frozen shoulder). we will apply interventions by this way For group A KT (kinesiology taping) will be applied on frozen shoulder patients by a professional physiotherapist or certified physiotherapist according to their pain pattern in muscles (supraspinatus, infraspinatus, teres minor, deltoid, subscapularis) with conventional physiotherapy of frozen shoulder also continues on 15 patients (group A). KT will apply twice a week for 8 weeks. We can check the results of our intervention every week by using variable tools or outcome measures, measuring pain by VAD (visual analog scale) and quality of life in the frozen shoulder by SPADI (shoulder pain and disability index) every week. And for group B Dry needling with conventional physical therapy.

DETAILED DESCRIPTION:
"Randomized control trial is our study design, we will make 2 groups group A ( 15 patients of frozen shoulder) and Group B (15 patients of frozen shoulder). we will apply interventions by this way For group A KT (kinesiology taping) will be applied on frozen shoulder patients by a professional physiotherapist or certified physiotherapist according to their pain pattern in muscles (supraspinatus, infraspinatus, teres minor, deltoid, subscapularis) with conventional physiotherapy of frozen shoulder also continues on 15 patients (group A). KT will apply twice a week for 8 weeks. We can check the results of our intervention every week by using variable tools or outcome measures, measuring pain by VAD (visual analog scale) and quality of life in the frozen shoulder by SPADI (shoulder pain and disability index) every week. And for group B Dry needling with conventional physical therapy.

DN ( dry needling) is applied on trigger points in the muscles (at a time two muscles) muscles would be supraspinatus, infraspinatus, teres minor, subscapularis, deltoid, and also used in myofascial pain around the shoulder joint combine with conventional physical therapy. Applying to the other 15 patients group B Needles with lengths of 25 to 40mm and widths of 0.25mm will be used. Each needle will be used once. 1 to 2 minutes for each trigger point. DN will apply twice a week for 8 weeks. We can check the results of our intervention every week by using variable tools or outcome measures, measuring pain by VAD (visual analog scale) and quality of life in the frozen shoulder by SPADI (shoulder pain and disability index) every week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with frozen shoulder
* Pain in the shoulder for at least 2 months before
* Available trigger points for at least one muscle around the shoulder joint (supraspinatus, deltoid, infraspinatus, teres minor, and subscapularis).
* Limited range of motion in internal rotation, external rotation, and abduction.

Exclusion Criteria:

* Patients with a history of allergy, pregnancy, or lactation period are excluded from the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
VAS | 6 Month
  visual Analog scale
SPADI | 6 Months
  shoulder pain and disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Pain away Physical Therapy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No